CLINICAL TRIAL: NCT03967730
Title: Sonodynamic Therapy in the Treatment of Perivascular Adipose Tissue on Patients With PAD and Claudication
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: COVID-19
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ye Tian PVAT
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2019-05

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sonodynamic therapy(SDT) (Experimental): Sonodynamic therapy(SDT) treatment is the combination of sonosensitizer administration and target atherosclerotic lesions ultrasound exposure.
  Interventions: Combination Product: Sonodynamic therapy(SDT)

INTERVENTIONS:
Combination Product: Sonodynamic therapy(SDT) — Sonodynamic Therapy (SDT) Sinoporphyrin Sodium (DVDMS) as sonosensitizer, is dissolved in 0.9% sodium solution for following skin test and intravenous injection. 0.01mg/ml DVDMS solution (0.1ml) is prepared for skin test followed by 0.04 mg/ml DVDMS solution intravenous injection(0.2mg/kg).The target atherosclerotic lesions are marked on the corresponding skin with ultrasound guidance and underwent ultrasound exposure after 4 hours incubation. The therapeutic ultrasonic transducer is fixed to the marked skin site for 15 min of each lesion. Ultrasound parameters included intensity of 2.1W/cm2 for each lesion, resonance frequency: 1.0 MHz and duty factor: 30%.

SUMMARY:
The purpose of this trial is to evaluate the safety and efficacy of sonodynamic therapy (SDT) in reducing the inflammation of perivascular adipose tissue and increasing peak walking time (PWT) among peripheral artery disease (PAD) patients with symptom of intermittent claudication.

DETAILED DESCRIPTION:
Atherosclerotic lower extremity PAD affects the living quality of more than 20 million people in the world. PAD is associated with a major decline in functional status and claudication is the most evident symptom. Current claudication therapies reveal significant limitations. Pharmacotherapy and exercise are recommended in 2016 AHA/ACC Guideline on the management of lower extremity PAD patients with claudication. However, they may not achieve an ideal clinical therapeutic effect. Furthermore, endovascular procedure may not be feasible, durable or cost-effective, especially in femoropopliteal arteries.

The aim of this trial is to verify the hypothesis that SDT can reduce the inflammation of PVAT and improve PWT among PAD patients with symptom of intermittent claudication.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-80 years
* Patients with atherosclerotic peripheral artery disease with symptoms of moderate to severe intermittent claudication (defined as ability to walk at least 2, but not more than 11 minutes on a graded treadmill test using the Gardner protocol)
* Femoral popliteal artery with 50% stenosis by ultrasound
* Stable use of low to moderate dose statin and the permitted statin drugs/ doses: atorvastatin 20 mg, simvastatin 40 mg, rosuvastatin 10 mg, pravastatin, 40 mg, fluvastatin 80 mg or lovastatin 40 mg for at least 6 weeks prior to screening
* Written informed consent

Exclusion Criteria:

* Severe aorto-iliac arteries stenosis or occlusion documented by noninvasive and invasive anatomic assessments
* Critical limb ischemia or other comorbid conditions that limit walking ability
* Non-atherosclerotic peripheral artery stenosis
* Active systemic inflammatory disease or have an infectious disease within 1 month prior to enrollment
* Systemic disorders such as hepatic, renal, hematologic, and malignant disease
* Allergic to contrast media with iodine
* Contraindication to CTA
* Allergic to DVDMS
* Diagnosis of porphyria
* Pregnant women and nursing mothers
* Patient who is attending other clinical trial

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-20 (Estimated); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in PVAT Density, as assessed by CTA | Measured at Baseline, 1, 3 months
  The changes in CT attenuation (HU) of perivascular adipose tissue(PVAT) as assessed by CTA.

SECONDARY OUTCOMES:
PWT change, mins | Measured at Baseline, 1, 3 months
  Changes from baseline peak walking time (PWT) at 1 month is assessed by graded treadmill test (Gardner protocol). The patient continues the test until walking can no longer be tolerated because of claudication symptoms.
Change in peak flow velocity, as assessed by doppler ultrasound | Measured at Baseline, 1, 3 months
  The changes of the systolic and diastolic peak flow velocity of the affected segments by doppler ultrasound.
Incidence of adverse events | Measured at Baseline, 1, 3 months
  Allergic to sunshine,hepatic or renal dysfunction,thyroid dysfunction
Plasma adipokines level | Measured at Baseline, 1, 3 months
  Including adiponectin, vaspin, apelin, leptin, visfatin, resistin and FABP
Plasma inflammation cytokine level | Measured at Baseline, 1, 3 months
  Including Interleukin-6(IL-6), IL-10, IL-1β, TGF-α, CRP, EGF, glutathione(GSH) and TGSH.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Tian, MD,PHD, Principal Investigator — First Affiliated Hospital of Harbin Medical University